CLINICAL TRIAL: NCT07206368
Title: Health Promotion With Targeted Exercise Intervention for Decreasing Fall Risk and Inactivity in Aging Veterans With Obesity and Signs of Sarcopenia
Acronym: ENHANCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRD8-002-24W; 1IK2RD000462 (Other Grant/Funding Number: Veterans Affairs Rehabilitation RDT Service)
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Falls; Sarcopenia; Obesity
Keywords: fall
MeSH Terms: conditions — Sarcopenia; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EX + EDU (Experimental): Participation in a live virtual fall-prevention exercise intervention plus a health promotion education program.
  Interventions: Other: Fall prevention exercise; Other: Health promotion education
- EDU (Active Comparator): Participation in a live virtual health promotion education program alone.
  Interventions: Other: Health promotion education

INTERVENTIONS:
Other: Fall prevention exercise — Participants will attend a virtual exercise-based group fall prevention class that focuses on movement and obstacle negotiation 3 times per week for 3 months.
  Other Names: EX
  Arms: EX + EDU
Other: Health promotion education — Participants will attend a virtual group health promotion education class that focuses on reasons to maintain a healthy lifestyle and local resources to support them in this. The sessions will take place 1 time per week for 3 months.
  Other Names: EDU

SUMMARY:
Falls are a major health risk for older Veterans, especially those with both obesity and low muscle mass or strength (sarcopenia), which together increase the chances of falling and losing independence. Many older Veterans have difficulty staying active and often lack information about how to safely exercise. While current guidelines focus mostly on weight loss, losing weight alone can weaken muscles and bones, which may actually raise the risk of falls and injuries. This study is testing the benefits of a virtual group exercise program combined with health education. The goal is to find out if exercise combined with health education is better at lowering fall risk and improving daily activity than health education alone for Veterans with obesity and signs of sarcopenia.

DETAILED DESCRIPTION:
Veterans with age-related declines in muscle mass and function, known as sarcopenia, are more likely to experience a fall, functional decline, and have higher mortality risk. Experiencing falls and limited functional mobility related to sarcopenia contributes to poor overall health, limited community participation, and loneliness, especially for Veterans with obesity. This group is uniquely vulnerable, as traditional weight-loss focused interventions may worsen muscle and bone loss, paradoxically increasing fall and injury risk. There is an urgent need to identify a feasible and efficacious intervention to address functional limitation and fall risk in aging Veterans with obesity and sarcopenia which does not further compromise their health.

This project departs from the traditional weight-loss approach for older Veterans with obesity by prioritizing functional health and fall risk reduction through targeted exercise and health education, specifically for those with sarcopenia. The intervention leverages a live, virtual group format to overcome mobility and access barriers, integrates wearable sensors for precise outcome measurement, and addresses both physical and behavioral aspects of fall prevention in a scalable, Veteran-centered design. The project addresses key knowledge gaps including: the lack of tailored fall prevention strategies for older Veterans with both obesity and sarcopenia; limited evidence on whether exercise interventions are superior to health education alone in this population; and uncertainties about the best ways to preserve muscle quality and reduce disability without compromising functional health through traditional weight-loss approaches. It also explores how virtual, group-based delivery can overcome access barriers for at-risk Veterans. The investigators will address these knowledge gaps through the following aims:

Aim 1: Compare the effects of a targeted exercise-based fall prevention intervention plus health promotion education program vs. health promotion education alone on clinical measures of fall risk and dysmobility. The investigators hypothesize Veterans participating in the combined exercise and health education program will show greater reductions in fall risk (primary outcome: Four Square Step Test (FSST)) compared to those receiving education alone.

Aim 2: Determine if combined exercise and health education and/or health promotion education alone result in physical activity changes indicative of greater ability to engage/engagement in community mobility. The investigators hypothesize Veterans participating in combined exercise and health education and those receiving health promotion education alone will show increased community mobility abilities evidenced by improved physical activity engagement (primary outcome: weekly minutes of moderate-vigorous physical activity), as measured through accelerometry. Those in combined exercise and health education are expected to have greater improvements compared to those in health promotion education alone.

Aim 3: Determine if combined exercise and health education and/or health promotion education alone result in changes to lower extremity muscle quality. The investigators hypothesize Veterans participating in combined exercise and health education will demonstrate improvements in functional muscle quality (primary outcome: knee extension strength) which are not expected to be observed for those in health promotion education alone.

This study will inform tailored strategies for fall prevention in aging Veterans with obesity and sarcopenia, supporting updated clinical practice guidelines that go beyond weight loss. It leverages innovative, scalable, Veteran-centered virtual interventions designed to optimize independence for Veterans at high risk for falls.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* 55 years or older
* VA primary care provider
* Enrolled in the VA Maryland Health Care System for health care
* Body mass index between and including 30 - 40 kg/m^2
* Showing signs of sarcopenia

Exclusion Criteria:

* Poorly controlled hypertensin
* Home oxygen use
* Contraindications to exercise or resistance exercise
* Significant cognitive impairment
* Other medical condition precluding patient participation in this study per the medical judgement of the study team

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Balance | 3 months
  The four-square step test will be used as a measure of balance. The change in amount of time it takes to complete the four-square step test is compared pre and post intervention
Physical activity | 3 months
  Weekly minutes of moderate-vigorous physical activity will be used as a measure of physical activity. The change in amount of weekly minutes is compared pre to post intervention.
Knee extension strength | 3 months
  A measure of the maximal isometric muscle strength produced in knee extensor muscles will be assessed with a handheld dynamometer device. Pre and post intervention levels will be compared.

SECONDARY OUTCOMES:
Mobility | 3 months
  The timed up and go will be used as a measure of mobility. The change in amount of time it takes to complete the timed up and go test is compared pre to post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Julie S Rekant, DPT PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No